CLINICAL TRIAL: NCT02535286
Title: Phase I Study of Ublituximab and Umbralisib in Combination With Targeted Immunotherapy in Patients With Relapsed-refractory Chronic Lymphocytic Leukemia (CLL) or Richter's Transformation (RT) of CLL
Brief Title: Study of Immunotherapy in Combination With Ublituximab and Umbralisib in Patients With Relapsed-refractory CLL or Richter's Transformation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-UPCC-108
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Chronic Lymphocytic Leukemia; Richter Syndrome
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — umbralisib; ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TG-1501 + Ublituximab + Umbralisib (Experimental): Ublituximab at a fixed IV infusion dose Days 1, 8 and 15 followed by maintenance infusions Umbralisib oral daily dose TG-1501 IV infusion at scheduled intervals
  Interventions: Drug: Umbralisib; Biological: ublituximab; Biological: TG-1501

INTERVENTIONS:
Drug: Umbralisib — A once daily oral agent
  Other Names: TGR-1202
Biological: ublituximab — IV anti-CD20 monoclonal antibody
  Other Names: TG-1101
Biological: TG-1501 — IV immunotherapy for cancer

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of targeted immunotherapy in combination with ublituximab and umbralisib, in patients with advanced CLL or Richter's Transformation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of B-cell Chronic Lymphocytic Leukemia or Richter's Transformation
* Refractory to or relapsed after at least 1 prior treatment regimen
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 14 days
* Known hepatitis B virus, hepatitis C virus or HIV infection
* Active autoimmune disorder (with the exception of autoimmune hemolytic anemia or ITP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-09-18 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Determine Acceptable Adverse Events That Are Related to Treatment | 6 months of therapy
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  The overall response rate (ORR) in patients with CLL and Richter's Transformation treated with Ublituximab in combination with Umbralisib and Targeted Immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R. Mato, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Seattle, Washington